CLINICAL TRIAL: NCT03218514
Title: Evaluating Body Size Descriptors on Peak Anti-Xa Levels in Bariatric Surgery Obese Patients Receiving Low Molecular Weight Heparin Fixed Doses
Brief Title: Venous Thromboprophylaxis in Bariatric Surgery
Acronym: OBSUD
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-07
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: Obesity; Venous thromboembolism; Heparin, Low-Molecular-Weight; Body Composition; Glomerular filtration rate; Bariatric Surgery
MeSH Terms: conditions — Obesity; Venous Thromboembolism | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Drug: Dalteparin

SUMMARY:
The main aim of this study is to compare the influence of total body-weight (TBW), lean body-weight (LBW), ideal body-weight (IBW) or Body Mass Index (BMI) on peak anti-Xa levels at steady-state in bariatric surgery (BS) morbidly obese patients receiving a fixed double dose of dalteparin (5000 IU subcutaneously, twice daily a day) for venous thromboembolism (VTE) prevention. Secondary aims of this study are to identify which body size descriptors (BSD) has the greatest impact and could further be explored for an adjusted low molecular weight heparin (LMWH) dosing algorithm for achieving optimal VTE prevention in BS severely obese patients.

DETAILED DESCRIPTION:
Severely obese patients undergoing bariatric surgery (BS) are at increased risk for venous thromboembolism (VTE). How standard LMWH regimen should be adapted to provide both sufficient efficacy and safety in this setting is unclear. The aim of this study is to compare the influence of four BSD on peak anti-Xa levels in BS obese patients receiving high LMWH fixed doses to identify which one had the greatest impact and could further be proposed in LMWH-based thromboprophylaxis dosing algorithms.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years old
* BMI ≥ 40 Kg/m² or BMI ≥ 35 Kg/m² with at least one or more obesity-related co-morbidities ( including type II diabetes (T2DM), hypertension, obstructive sleep apnea (OSA), non-alcoholic fatty liver disease, severe osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease)
* scheduled for sleeve gastrectomy (SG) or gastric bypass procedure (GBP)
* informed consent

Exclusion Criteria:

* anticoagulant administration within 48 hours preceding surgery
* on-going antiplatelet therapy
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose peak plasma anti-Xa levels is in the prophylactic ranges | at least two days after thromboprophylaxis initiation
  Proportion of patients whose peak plasma anti-Xa levels is in the prophylactic ranges.The target range for prophylactic anti-Xa levels is defined as 0.2 to 0.5 IU/ml

SECONDARY OUTCOMES:
Proportion of patients with symptomatic VTE | 3 months
  Proportion of patients with symptomatic VTE
Proportion of patients with major bleeding | 3 months
  Proportion of patients with major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Gaborit, Principal Investigator — Inserm U1062, Inra U1260, Aix Marseille Université, Faculté de Médecine, Assistance Publique - Hôpitaux de Marseille

REFERENCES:
- [Result] Gaborit B, Aron-Wisnewsky J, Salem JE, Bege T, Frere C. Pharmacologic Venous Thromboprophylaxis After Bariatric Surgery: Burning Questions Regarding Doses, Duration, and Strategy. Ann Surg. 2018 Dec;268(6):e51-e52. doi: 10.1097/SLA.0000000000002536. No abstract available. PMID 28938272
- [Result] Gaborit B, Moulin PA, Bege T, Boullu S, Vincentelli C, Emungania O, Morange PE, Berdah S, Salem JE, Dutour A, Frere C. Lean body weight is the best scale for venous thromboprophylaxis algorithm in severely obese patients undergoing bariatric surgery. Pharmacol Res. 2018 May;131:211-217. doi: 10.1016/j.phrs.2018.02.012. Epub 2018 Feb 13. PMID 29452290